CLINICAL TRIAL: NCT04908150
Title: A Core Training Protocol Achieves Improvements in Function, Motor Control and Endurance Strength Compared to a Traditional Abdomen Exercise Protocol: a Randomised Controlled Trial.
Brief Title: Core Training Protocol vs Traditional Abdomen Exercise Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Manuel González-Sánchez (Other)
Responsible Party: Sponsor-Investigator, Dr. Manuel González-Sánchez, Principal Investigator, University of Malaga
Organization: University of Malaga (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111-2020
Record Dates: First submitted 2021-05-21; First posted 2021-06-01 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Functional Performance; Resistance Training; Exercise
Keywords: prevention; core; accelerometer; functional
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core Group (Experimental): The Core Group carried out core stability exercises. Their training consisted of the following exercises: bridge, Klapp, front plank and lateral plank
  Interventions: Other: Core training
- Abdominal Group (Active Comparator): The Abdominal Group performed traditional exercises: trunk flexion or abdominal crunch, trunk extensions, lower abdominals with hip lifts and crunch with crossed legs
  Interventions: Other: Core training

INTERVENTIONS:
Other: Core training — A total of 12 sessions were carried out, which lasted for 4 weeks, with a frequency of 3 sessions/ week. The duration of each session was 11 minutes 30 seconds. The working time of each exercise was 30 seconds with a 5 seconds rest between exercises, meaning that each exercise cycle lasted for 2.50 seconds. Three exercise cycles were performed with a 90 seconds rest between each one of them

SUMMARY:
The main objective of this study is to analyse the effectiveness of core stability exercises to increase motor control, function and resistance strength of the abdominal muscles, compared to a traditional abdominal and trunk exercise program in semi-professionals soccer players

DETAILED DESCRIPTION:
The 51 participants were semi-professional soccer player and were divided into two different groups using a computer system: the CORE-group or ABDOMINALS-group. Four weeks of training were developed. Outcome variables: Back extension test; Flexion endurance test; FMS; functional movement screen; lateral muscle test right; lateral muscle test left. Kinematic variables were recorded during the test using an accelerometer. A comparison intra-group and intergroup were developed.

ELIGIBILITY:
Inclusion Criteria:

* semi-professional soccer player

Exclusion Criteria:

* Participants who have suffered a musculoskeletal pathology in the lower limbs and/or having undergone some surgical intervention in the prior year were excluded

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Functional Movement Screen | 5 minutes
  motor control and functionality in movement
McGill test | 5 minutes
  resistance strength of the abdominal muscle

CONTACTS AND LOCATIONS:
Locations (1):
- Manuel Gonzalez-Sanchez, Málaga, Spain

IPD SHARING:
Plan to Share IPD: Yes
publication in a scientific journal
Supporting Information: Study Protocol, SAP
Time Frame: one month
Access Criteria: open access